CLINICAL TRIAL: NCT06382428
Title: Comparison of the Effects of Pelvic Floor Muscle Training Applied With the Telerehabilitation Method and Supervised in the Postpartum Period on Pelvic Floor Muscle Function, Pelvic Floor Symptoms and Quality of Life
Brief Title: The Effects of Pelvic Floor Muscle Training Applied With the Telerehabilitation Method in the Postpartum Period
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Tinaztepe University (Other)
Collaborators: Biruni University (Other); Yeditepe University (Other); Fenerbahce University (Other)
Responsible Party: Principal Investigator, Damla Korkmaz Dayican, Lecturer, Izmir Tinaztepe University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: T-DAYICAN-002
Record Dates: First submitted 2024-04-17; First posted 2024-04-24 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Pelvic Floor Disorders; Postpartum Disorder; Quality of Life; Mothers
Keywords: Pelvic floor muscle training; Postpartum; Telerehabilitation; Quality of Life
MeSH Terms: conditions — Pelvic Floor Disorders; Puerperal Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TR-PFMT group (Experimental): In the TR-PFMT group, the PFMT program was carried out via a synchronous online platform (Skype™ program). Participants were asked to install Skype™ software on their personal computers or phones and create a personal account. In the first evaluation session, participants were taught how to use the hardware and software. Additionally, they were asked to place their cameras at an average distance of 1-1.5 meters so that their entire body could be seen. At the beginning of each session, they were informed that their information was kept confidential and their audio and video images would not be shared with another person.
  Interventions: Other: Pelvic floor muscle training
- S-PFMT group (Active Comparator): In the S-PFMT group, the PFMT program was conducted as a face-to-face session in groups of 4 people.
  Interventions: Other: Pelvic floor muscle training

INTERVENTIONS:
Other: Pelvic floor muscle training — The PFMT program was carried out for 45-50 minutes, 2 days a week for 8 weeks, by two physiotherapists specialized experienced in the pelvic floor. The program consisted of education, diaphragm breathing exercises, pelvic mobility exercises, exercises to strengthen and stretch the pelvic floor muscles and other muscles related to the pelvis. In addition, the participants were expected to do the same exercises at home 2 days a week.

SUMMARY:
Pelvic floor muscle training (PFMT) is routinely recommended to treat and prevent pelvic floor symptoms in the postpartum period. However, due to the high cost, remoteness of the location, and responsibilities of the baby, women cannot participate in PFMT whenever and wherever they want. Telerehabilitation (TR) may be an effective method to facilitate women's access to PFMT. Therefore, our study aims to compare the short and medium-term effects of PFMT applied with the TR method on pelvic floor symptoms, symptom-related quality of life and pelvic floor muscle function with supervised PFMT. This randomized controlled study was conducted at Yeditepe University Hospital Bağdat Street Polyclinic Pelvic Floor Center and online synchronous platform on women aged 18-35 and between the 6th and 8th weeks postpartum. Participants were randomly assigned to the synchronized PFMT performed with the telerehabilitation method (TR-PFMT) group and the supervised PFMT (S-PFMT) group. The same PFMT program was carried out in both groups for 45-50 minutes, 2 days a week for 8 weeks, by two physiotherapists specialized experienced in the pelvic floor. The program was carried out via a synchronous online platform (Skype™ program) in the TR-PFMT group, and as a face-to-face session in the S-PFMT group. Participants' pelvic floor symptoms were evaluated with the Pelvic Floor Distress Inventory-20 (PFDI-20), symptom-related quality of life was evaluated with the Pelvic Floor Impact Questionnaire-7 (PFIQ-7), and pelvic floor muscle function was evaluated with superficial electromyography. Evaluations were made 3 times in total: before the exercise program, after the exercise program and at the 8th week after the exercise program (6th month postpartum).

ELIGIBILITY:
Inclusion Criteria:

* Being a woman between 18-35 years old
* Between the 6th and 8th weeks postpartum
* Native Turkish
* Having the appropriate technological infrastructure to participate in an exercise session via the Internet (for the TR-PFMT group)

Exclusion Criteria:

* Number of births >2
* The week of pregnancy <32
* Having a history of 3rd and 4th-degree perineal tears
* Cesarean birth
* Inability to contract the pelvic floor muscle (pelvic floor muscle strength ≤2 according to the Modified Oxford Scale)
* The electromyography values of the abdominal muscles or hip adductors during contraction of the pelvic floor muscles are more than 10 microvolts
* The presence of neurological, orthopedic, psychiatric, hematological or cardiovascular disease that would prevent PFMT as questioned by the gynecologist
* Body mass index ≥ 25 kg/m²
* The presence of active urinary tract or vaginal infection in the last week

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2022-12-30 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
Pelvic Floor Distress Inventory-20 to measure the total pelvic floor symptoms | pre-intervention; immediately after the intervention
  It was used to assess the severity of the pelvic floor symptoms such as pelvic organ prolapse, colorectal-anal, and urinary symptoms. It consists of 20 questions and three subdimensions: Pelvic Organ Prolapse Distress Inventory-6, Colorectal-Anal Distress Inventory-8, and Urinary Distress Inventory-6. Each subdimension is averaged and multiplied by 25 to convert the score of the scale to a number out of 100. The score of the subdimension ranges from 0 to 100 and the total score ranges from 0 to 300. A higher score on the scale indicates greater severity of the complaints.
Pelvic Floor Distress Inventory-20 to measure the pelvic organ prolapse symptoms | pre-intervention; immediately after the intervention
  It was used to assess the severity of the pelvic floor symptoms such as pelvic organ prolapse, colorectal-anal, and urinary symptoms. It consists of 20 questions and three subdimensions: Pelvic Organ Prolapse Distress Inventory-6, Colorectal-Anal Distress Inventory-8, and Urinary Distress Inventory-6. Each subdimension is averaged and multiplied by 25 to convert the score of the scale to a number out of 100. The score of the subdimension ranges from 0 to 100 and the total score ranges from 0 to 300. A higher score on the scale indicates greater severity of the complaints.
Pelvic Floor Distress Inventory-20 to measure the colorectal-anal symptoms | pre-intervention; immediately after the intervention
  It was used to assess the severity of the pelvic floor symptoms such as pelvic organ prolapse, colorectal-anal, and urinary symptoms. It consists of 20 questions and three subdimensions: Pelvic Organ Prolapse Distress Inventory-6, Colorectal-Anal Distress Inventory-8, and Urinary Distress Inventory-6. Each subdimension is averaged and multiplied by 25 to convert the score of the scale to a number out of 100. The score of the subdimension ranges from 0 to 100 and the total score ranges from 0 to 300. A higher score on the scale indicates greater severity of the complaints.
Pelvic Floor Distress Inventory-20 to measure the urinary symptoms | pre-intervention; immediately after the intervention
  It was used to assess the severity of the pelvic floor symptoms such as pelvic organ prolapse, colorectal-anal, and urinary symptoms. It consists of 20 questions and three subdimensions: Pelvic Organ Prolapse Distress Inventory-6, Colorectal-Anal Distress Inventory-8, and Urinary Distress Inventory-6. Each subdimension is averaged and multiplied by 25 to convert the score of the scale to a number out of 100. The score of the subdimension ranges from 0 to 100 and the total score ranges from 0 to 300. A higher score on the scale indicates greater severity of the complaints.
Pelvic Floor Impact Questionnaire-7 to measure the total pelvic floor symptoms related quality of life | pre-intervention; immediately after the intervention
  It was used to evaluate the impact of pelvic floor symptoms on quality of life. It consists of 21 questions and three subdimensions: Urinary Impact Questionnaire-7, Colorectal-Anal Impact Questionnaire-7, and Pelvic Organ Prolapse Impact Questionnaire-7. It is calculated by taking the average of each subdimension and multiplying it by 100/3 to convert the score of the scale into a 100-point system. The score of the subdimension ranges from 0 to 100 and the total score ranges from 0 to 300. A high score indicates that the pelvic floor symptoms negatively affect quality of life.
Pelvic Floor Impact Questionnaire-7 to measure the pelvic organ prolapse symptoms related quality of life | pre-intervention; immediately after the intervention
  It was used to evaluate the impact of pelvic floor symptoms on quality of life. It consists of 21 questions and three subdimensions: Urinary Impact Questionnaire-7, Colorectal-Anal Impact Questionnaire-7, and Pelvic Organ Prolapse Impact Questionnaire-7. It is calculated by taking the average of each subdimension and multiplying it by 100/3 to convert the score of the scale into a 100-point system. The score of the subdimension ranges from 0 to 100 and the total score ranges from 0 to 300. A high score indicates that the pelvic floor symptoms negatively affect quality of life.
Pelvic Floor Impact Questionnaire-7 to measure the colorectal-anal symptoms related quality of life | pre-intervention; immediately after the intervention
  It was used to evaluate the impact of pelvic floor symptoms on quality of life. It consists of 21 questions and three subdimensions: Urinary Impact Questionnaire-7, Colorectal-Anal Impact Questionnaire-7, and Pelvic Organ Prolapse Impact Questionnaire-7. It is calculated by taking the average of each subdimension and multiplying it by 100/3 to convert the score of the scale into a 100-point system. The score of the subdimension ranges from 0 to 100 and the total score ranges from 0 to 300. A high score indicates that the pelvic floor symptoms negatively affect quality of life.
Pelvic Floor Impact Questionnaire-7 to measure the urinary symptoms related quality of life | pre-intervention; immediately after the intervention
  It was used to evaluate the impact of pelvic floor symptoms on quality of life. It consists of 21 questions and three subdimensions: Urinary Impact Questionnaire-7, Colorectal-Anal Impact Questionnaire-7, and Pelvic Organ Prolapse Impact Questionnaire-7. It is calculated by taking the average of each subdimension and multiplying it by 100/3 to convert the score of the scale into a 100-point system. The score of the subdimension ranges from 0 to 100 and the total score ranges from 0 to 300. A high score indicates that the pelvic floor symptoms negatively affect quality of life.
Surface electromyography (EMG) to measure the pre-basal activity of the pelvic floor muscles | pre-intervention; immediately after the intervention
  The NeuroTract Myoplus 2 PRO (Verity Medical LTD., UK) brand EMG device was used to evaluate pelvic floor muscle function. EMG activities of the pelvic floor muscles were recorded with disposable 3.2 x 3.2 cm superficial electrodes. Bipolar electrodes were placed on the right and left sides of the perineal body (3-9 o'clock), and the monopolar reference electrode was placed on the right spina iliac anterior superior. Measurements were performed in the supine position during voluntary relaxation and voluntary contraction of the pelvic floor muscles. The Glazer Protocol, which is a valid and reliable method to evaluate pelvic floor muscle function, was used. According to this protocol, Pre-baseline rest activity, phasic activity, tonic activity, endurance activity and post-baseline rest activity of the pelvic floor muscles were evaluated. EMG activities were automatically recorded by the device.
Surface electromyography (EMG) to measure the phasic activity of the pelvic floor muscles | pre-intervention; immediately after the intervention
  The NeuroTract Myoplus 2 PRO (Verity Medical LTD., UK) brand EMG device was used to evaluate pelvic floor muscle function. EMG activities of the pelvic floor muscles were recorded with disposable 3.2 x 3.2 cm superficial electrodes. Bipolar electrodes were placed on the right and left sides of the perineal body (3-9 o'clock), and the monopolar reference electrode was placed on the right spina iliac anterior superior. Measurements were performed in the supine position during voluntary relaxation and voluntary contraction of the pelvic floor muscles. The Glazer Protocol, which is a valid and reliable method to evaluate pelvic floor muscle function, was used. According to this protocol, Pre-baseline rest activity, phasic activity, tonic activity, endurance activity and post-baseline rest activity of the pelvic floor muscles were evaluated. EMG activities were automatically recorded by the device.
Surface electromyography (EMG) to measure the tonic activity of the pelvic floor muscles | pre-intervention; immediately after the intervention
  The NeuroTract Myoplus 2 PRO (Verity Medical LTD., UK) brand EMG device was used to evaluate pelvic floor muscle function. EMG activities of the pelvic floor muscles were recorded with disposable 3.2 x 3.2 cm superficial electrodes. Bipolar electrodes were placed on the right and left sides of the perineal body (3-9 o'clock), and the monopolar reference electrode was placed on the right spina iliac anterior superior. Measurements were performed in the supine position during voluntary relaxation and voluntary contraction of the pelvic floor muscles. The Glazer Protocol, which is a valid and reliable method to evaluate pelvic floor muscle function, was used. According to this protocol, Pre-baseline rest activity, phasic activity, tonic activity, endurance activity and post-baseline rest activity of the pelvic floor muscles were evaluated. EMG activities were automatically recorded by the device.
Surface electromyography (EMG) to measure the endurance activity of the pelvic floor muscles | pre-intervention; immediately after the intervention
  The NeuroTract Myoplus 2 PRO (Verity Medical LTD., UK) brand EMG device was used to evaluate pelvic floor muscle function. EMG activities of the pelvic floor muscles were recorded with disposable 3.2 x 3.2 cm superficial electrodes. Bipolar electrodes were placed on the right and left sides of the perineal body (3-9 o'clock), and the monopolar reference electrode was placed on the right spina iliac anterior superior. Measurements were performed in the supine position during voluntary relaxation and voluntary contraction of the pelvic floor muscles. The Glazer Protocol, which is a valid and reliable method to evaluate pelvic floor muscle function, was used. According to this protocol, Pre-baseline rest activity, phasic activity, tonic activity, endurance activity and post-baseline rest activity of the pelvic floor muscles were evaluated. EMG activities were automatically recorded by the device.
Surface electromyography (EMG) to measure the post-baseline rest activity of the pelvic floor muscles | pre-intervention; immediately after the intervention
  The NeuroTract Myoplus 2 PRO (Verity Medical LTD., UK) brand EMG device was used to evaluate pelvic floor muscle function. EMG activities of the pelvic floor muscles were recorded with disposable 3.2 x 3.2 cm superficial electrodes. Bipolar electrodes were placed on the right and left sides of the perineal body (3-9 o'clock), and the monopolar reference electrode was placed on the right spina iliac anterior superior. Measurements were performed in the supine position during voluntary relaxation and voluntary contraction of the pelvic floor muscles. The Glazer Protocol, which is a valid and reliable method to evaluate pelvic floor muscle function, was used. According to this protocol, Pre-baseline rest activity, phasic activity, tonic activity, endurance activity and post-baseline rest activity of the pelvic floor muscles were evaluated. EMG activities were automatically recorded by the device.

CONTACTS AND LOCATIONS:
Overall Officials: Arzu Razak Özdinçler, PT, PhD, Prof., Study Director — Fenerbahçe University; Damla Korkmaz Dayıcan, PT, PhD (c), Principal Investigator — İzmir Tınaztepe University; Burçin Özyürek, PT, PhD (c), Principal Investigator — Yeditepe University
Locations (1):
- Yeditepe University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No